CLINICAL TRIAL: NCT00504205
Title: Safety Study to Determine the Maximum Tolerated Dose, Pharmacokinetics and Pharmacodynamics of Oral MP470, a Multi-Targeted Tyrosine Kinase Inhibitor, in Patients With Solid Malignancies
Brief Title: MP470 in Treating Patients With Unresectable or Metastatic Solid Tumor or Lymphoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn as trial was never activated by SuperGen
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SUPERGEN-SGI-0470-01; CDR0000556524 (Registry Identifier: PDQ (Physician Data Query)); VPCCS-SGI-0470-01
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-04

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; intraocular lymphoma; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV small lymphocytic lymphoma; Waldenstrom macroglobulinemia; primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Waldenstrom Macroglobulinemia | interventions — amuvatinib; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: multitargeted receptor tyrosine kinase inhibitor MP470
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: positron emission tomography

SUMMARY:
RATIONALE: MP470 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This clinical trial is studying the side effects and best dose of MP470 in treating patients with unresectable or metastatic refractory solid tumor, Hodgkin's lymphoma, or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the maximum tolerated dose (MTD) and define the safety profile of multitargeted receptor tyrosine kinase inhibitor MP470 in humans.

Secondary

* Estimate the therapeutic response rate for patients receiving MP470.
* Define the human pharmacokinetic (PK) and pharmacodynamic (PD) profiles of MP470 capsules
* Evaluate PK-PD relationships.

OUTLINE: This is a multicenter study.

Patients receive oral multitargeted receptor tyrosine kinase inhibitor MP470 until the maximum tolerated dose is determined.

Pharmacokinetic and pharmacodynamic analyses are carried out to determine changes in phosphorylation of extracellular signal-regulated kinase (ERK), Rad51 expression, number of circulating tumor cells (CTCs), and tumor glucose metabolism measured by 2-[18F]fluoro-2-deoxyglucose positron emission tomography (FDG-PET).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histological or cytological diagnosis of unresectable or metastatic solid-tumor cancer that is refractory to standard therapies OR for which no standard therapy exists

  * Patients with refractory lymphoma (Hodgkin or non-Hodgkin) are also permitted to participate

Exclusion criteria:

* Active CNS metastases (primary brain tumors are permitted)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status ≥ 70%
* Hemoglobin ≥ 9 g/dL
* ANC ≥ 1.5 × 10^9/L
* Platelet count ≥ 100 × 10^9/L
* Total serum bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 2.5 × ULN (upper limit of normal for the clinical laboratory), but ≤ 5 × ULN is acceptable if due to hepatic metastases
* Serum albumin ≥ 2 g/dL
* Serum creatinine ≤ 2 mg/dL
* LVEF ≥ 50% on ECHO
* No significant abnormalities on the screening ECG (e.g., left bundle branch block, 3rd degree AV block, acute myocardial infarction or QTc interval > 450 msec)
* No history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia or family history of Long QT Syndrome)
* Able to swallow MP470 capsules
* Capable of fasting for 6 hours
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months following completion of study treatment

Exclusion criteria:

* Life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of oral MP470, or put the study outcomes at risk
* Any serious, uncontrolled active infection that requires systemic treatment
* History of significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, and/or myocardial infarction

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Recuperated from any prior surgical procedures including at least 4 weeks rest since a major surgery

Exclusion criteria:

* Patient has received any anticancer agent(s) within the past 3 weeks, including investigational agents, chemotherapy (6 weeks for nitrosoureas or mitomycin), immunotherapy, biologic, or hormonal therapy other than luteinizing hormone-releasing hormone (LHRH) agonists
* Patient has received radiation therapy within the past 4 weeks
* Patient has a grade 2 or more severe toxicity (other than alopecia) continuing from prior anticancer therapy
* Patient requires treatment with immunosuppressive agents other than corticosteroids that have been at stable doses for at least 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety
Response to treatment according to RECIST criteria
Pharmacodynamic assessments (e.g., changes in phosphorylation of ERK, Rad51 expression, number of CTCs, and tumor glucose metabolism measured by FDG-PET)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Berk, MD, Study Chair — Astex Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas